CLINICAL TRIAL: NCT02165722
Title: An Enhanced 4 Pillars Toolkit for Increasing Adolescent Immunization: A Randomized Controlled Cluster Trial in Pediatrics and Family Medicine
Brief Title: 4 Pillars Toolkit for Adolescent Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Pfizer (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Richard Zimmerman, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO13070205
Record Dates: First submitted 2014-06-13; First posted 2014-06-17 (Estimated); Results first posted 2018-07-30 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-07

CONDITIONS: Adolescent HPV Vaccine; Adolescent Influenza Vaccine
Keywords: Influenza; HPV; Tdap; MCV; vaccination; adolescents
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Toolkit (Experimental): 4 Pillars Toolkit
  Interventions: Behavioral: 4 Pillars Toolkit
- No Intervention: Standard practice (No Intervention): 11 Clinical Practices [control sites]

INTERVENTIONS:
Behavioral: 4 Pillars Toolkit — Behavioral: Pillar 1: Convenient Vaccination Services (e.g. use every visit [chronic and acute] as an opportunity to vaccinate; use express vaccination clinics and dedicated vaccination stations; use influenza vaccination as an opportunity to vaccinate for other vaccines).
  Behavioral: Pillar 2: Patient Notification (e.g. use electronic reminders and social media for vaccination reminders; use physician recommendations).
  Behavioral: Pillar 3: Enhanced Office Systems (e.g. implement Standing Order Programs; use EMR prompts; add vaccination status as a vital sign when rooming).
  Behavioral: Pillar 4: Motivation (e.g. establish an office Immunization Champion to track goal progress, aided by research team feedback).
  Arms: Intervention: Toolkit

SUMMARY:
The purpose of this study is to test whether or not the 4 Pillars Immunization Toolkit increases adolescent vaccination rates, particularly influenza and human papillomavirus (HPV) but also tetanus, diphtheria and pertussis (Tdap), and meningococcal conjugate (MCV) vaccination rates. The vaccines are all FDA licensed vaccines and to be used according to national guidelines. The investigators will conduct a randomized cluster trial of this toolkit in diverse primary care practices with electronic medical records (EMRs).

DETAILED DESCRIPTION:
This intervention is a stratified randomized cluster trial in about 22 diverse primary care practices. These practices will be randomly assigned to be intervention or control sites to test this 4 Pillars Immunization Toolkit intervention package of evidence-based techniques tailored to their practice structure and culture; the specialties are split between pediatric and family medicine practices.

.

ELIGIBILITY:
Inclusion Criteria:

* For clinical sites: inclusion criterion includes

  1. an appropriate adolescent population: e.g., adolescents aged 11 to 17 years
  2. currently using an EMR
  3. having and keeping immunization data within a EMR or registry.

Exclusion Criteria:

* For clinical sites: the exclusion criteria is consistent SOP use for the vaccines being studied or known much higher than average immunization rates.

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2013-09; Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard K Zimmerman, MD, MPH, MA, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, School of Medicine, Department of Family Medicine, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zimmerman RK, Moehling KK, Lin CJ, Zhang S, Raviotta JM, Reis EC, Humiston SG, Nowalk MP. Improving adolescent HPV vaccination in a randomized controlled cluster trial using the 4 Pillars practice Transformation Program. Vaccine. 2017 Jan 3;35(1):109-117. doi: 10.1016/j.vaccine.2016.11.018. Epub 2016 Nov 18. PMID 27876200
- [Derived] Zimmerman RK, Raviotta JM, Nowalk MP, Moehling KK, Reis EC, Humiston SG, Lin CJ. Using the 4 Pillars Practice Transformation Program to increase adolescent human papillomavirus, meningococcal, tetanus-diphtheria-pertussis and influenza vaccination. Vaccine. 2017 Oct 27;35(45):6180-6186. doi: 10.1016/j.vaccine.2017.09.039. Epub 2017 Sep 22. PMID 28947346

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cluster randomized trial where units reflect clinical practices enrolled. Numbers of participants who started and ended study reflect the longitudinal analytic data set of patients who had a visit during both the baseline and intervention periods.
Units Other Than Participants: clinics
Groups:
- Intervention Sites: 9 Clinical practices (intervention sites) used the 4 Pillars Toolkit to increase vaccination rates from baseline to end of year 1. Two practices dropped out of the intervention (11-2=9).
  Patients: Adolescents aged 11-17 years of age who had a visit during both the baseline (7/1/2013 to 6/30/2014) and intervention periods (7/1/2014 to 3/31/2015).
  The 4 Pillars Toolkit is built around 4 pillars which include evidence-based strategies to increase vaccination rates:
  Pillar 1: Convenient Vaccination Services
  Pillar 2: Patient Notification
  Pillar 3: Enhanced Office Systems
  Pillar 4: Motivation
- Control Sites: 11 Clinical Practices [control sites] were not actively intervened upon.
  Patients: Adolescents aged 11-17 years of age who had a visit during both the baseline (7/1/2013 to 6/30/2014) and intervention periods (7/1/2014 to 3/31/2015).
Period: Overall Study
Arm/Group | Intervention Sites | Control Sites
Started | 1971; 9 clinics | 2202; 11 clinics
Completed | 1971; 9 clinics (Started and completed participants reflect the longitudinal analytic data set of patients used) | 2202; 11 clinics (Started and completed participants reflect the longitudinal analytic data set of patients used)
Not Completed | 0; 0 clinics | 0; 0 clinics

BASELINE CHARACTERISTICS:
Groups:
- Intervention Sites: Clinical practices: 9 Clinical practices (intervention sites) used the 4 Pillars Toolkit to increase vaccination rates from baseline to end of year 1.
  Patients: Adolescents aged 11-17 years of age who had a visit during both the baseline (7/1/2013 to 6/30/2014) and intervention periods (7/1/2014 to 3/31/2015).
- Control Sites: Clinical practices: 11 Clinical Practices [control sites] were not actively intervened upon but continued their standard clinical practices regarding provision of vaccinations.
  Patients: Adolescents aged 11-17 years of age who had a visit during both the baseline (7/1/2013 to 6/30/2014) and intervention periods (7/1/2014 to 3/31/2015).
- Total: Total of all reporting groups
Arm/Group | Intervention Sites | Control Sites | Total
Number analyzed (Participants) | 4,942 | 5,919 | 10861
Age, Customized [Number; unit: percent of participants aged 11-13 years]
  percent of participants aged 11-13 years | 39.9 | 37.2 | 38.4
Sex/Gender, Customized [Number; unit: percent of female participants]
  percent of female participants | 49.6 | 51.1 | 50.3
Race/Ethnicity, Customized [Number; unit: percent of Non-white participants]
  percent of Non-white participants | 12.0 | 23.4 | 18.2
Commercial health insurance, % [Number; unit: percent of participants privt insurance] | 62.2 | 67.8 | 64.7

OUTCOME MEASURES:

1. Primary Outcome: Change in Percentage of Cumulative HPV Series Initiation Vaccination Rates for Adolescents 11-17 Years of Age
Description: Change in cumulative vaccination rates from baseline to end of year 1 for HPV series initiation (e.g., receipt of first dose of HPV vaccine) stratified by age 11-13 years and 14-17 years. Baseline period was 7/1/2013 to 6/30/2014. Intervention period was 7/1/2014 to 3/31/2015.
Time Frame: Baseline period to post-intervention
Population: HPV series initiation stratified by age of 11-13 years and 14-17 years of age. Baseline period was 7/1/2013 to 6/30/2014. Intervention period was 7/1/2014 to 3/31/2015.
Measure: Number; unit: percent change in vaccination rates
Groups:
- Intervention Group: HPV Series Initiation 11-13 Years of Age; Intervention Group: HPV Series Initiation 14-17 Years of Age: Practices: Represents 9 clinical practices
  Patients: Adolescents aged 11-17 years of age who had a visit during both the baseline (7/1/2013 to 6/30/2014) and intervention periods (7/1/2014 to 3/31/2015).
  Baseline period was 7/1/2013 to 6/30/2014. Intervention period was 7/1/2014 to 3/31/2015.
- Control Group: HPV Series Initiation 11-13 Years of Age; Control Group: HPV Series Initiation 14-17 Years of Age: Practices: Represents 11 clinical practices
  Patients: Adolescents aged 11-17 years of age who had a visit during both the baseline (7/1/2013 to 6/30/2014) and intervention periods (7/1/2014 to 3/31/2015).
  Baseline period was 7/1/2013 to 6/30/2014. Intervention period was 7/1/2014 to 3/31/2015.
Arm/Group | Intervention Group: HPV Series Initiation 11-13 Years of Age | Control Group: HPV Series Initiation 11-13 Years of Age | Intervention Group: HPV Series Initiation 14-17 Years of Age | Control Group: HPV Series Initiation 14-17 Years of Age
Number analyzed (Participants) | 1,971 | 2,202 | 2,971 | 3,717
percent change in vaccination rates | 13.7 | 10.1 | 7.8 | 5.7
Statistical Analysis 1: Comparison: Intervention Group: HPV Series Initiation 11-13 Years of Age vs Intervention Group: HPV Series Initiation 14-17 Years of Age; Test type: Other — Chi-square tests performed to test for differences in cumulative HPV series initiation vaccination rates from baseline to post-intervention; p < 0.001, Chi-squared — Statistical significance for two-sided tests was set at a type I error (alpha) equal to 0.05; Chi-square tests performed to test for differences in cumulative HPV series initiation vaccination rates from baseline to post-intervention
Statistical Analysis 2: Comparison: Control Group: HPV Series Initiation 11-13 Years of Age vs Control Group: HPV Series Initiation 14-17 Years of Age; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.001, Chi-squared — Statistical significance for two-sided tests was set at a type I error (alpha) equal to 0.05; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Intervention Group: HPV Series Initiation 11-13 Years of Age vs Control Group: HPV Series Initiation 11-13 Years of Age; Chi-square tests performed to test for differences in cumulative HPV series initiation vaccination rates from baseline to post-intervention between intervention and control clinics; Test type: Other — Chi-square tests performed to test for differences in cumulative HPV series initiation vaccination rates from baseline to post-intervention between intervention and control clinics; p < 0.001, Chi-squared — Statistical significance for two-sided tests was set at a type I error (alpha) equal to 0.05
Statistical Analysis 4: Comparison: Intervention Group: HPV Series Initiation 14-17 Years of Age vs Control Group: HPV Series Initiation 14-17 Years of Age; Test type: Other — [test comment as in outcome 1, analysis 3]; p < 0.001, Chi-squared — Statistical significance for two-sided tests was set at a type I error (alpha) equal to 0.05

2. Primary Outcome: Change in Percentage of Cumulative HPV Series Completion Vaccination Rates for Adolescents 11-17 Years of Age
Description: Change in cumulative vaccination rates from baseline to end of year 1 for HPV series completion (e.g., receipt of third dose of HPV vaccine) stratified by age 11-13 years and 14-17 years. Baseline period was 7/1/2013 to 6/30/2014. Intervention period was 7/1/2014 to 3/31/2015.
Time Frame: Baseline period to post-intervention
Measure: Number; unit: percent change in vaccination rates
Groups:
- Intervention Group: HPV Series Completion 11-13 Years of Age; Intervention Group: HPV Series Completion 14-17 Years of Age: Practices: Represents 9 clinical practices
  Patients: Adolescents aged 11-17 years of age who had a visit during both the baseline (7/1/2013 to 6/30/2014) and intervention periods (7/1/2014 to 3/31/2015).
  Baseline period was 7/1/2013 to 6/30/2014. Intervention period was 7/1/2014 to 3/31/2015.
- Control Group: HPV Series Completion 11-13 Years of Age; Control Group: HPV Series Completion 14-17 Years of Age: Practices: Represents 11 clinical practices
  Patients: Adolescents aged 11-17 years of age who had a visit during both the baseline (7/1/2013 to 6/30/2014) and intervention periods (7/1/2014 to 3/31/2015).
  Baseline period was 7/1/2013 to 6/30/2014. Intervention period was 7/1/2014 to 3/31/2015.
Arm/Group | Intervention Group: HPV Series Completion 11-13 Years of Age | Control Group: HPV Series Completion 11-13 Years of Age | Intervention Group: HPV Series Completion 14-17 Years of Age | Control Group: HPV Series Completion 14-17 Years of Age
Number analyzed (Participants) | 1,971 | 2,202 | 2,971 | 3,717
percent change in vaccination rates | 14.8 | 15.8 | 11.6 | 10.8
Statistical Analysis 1: Comparison: Intervention Group: HPV Series Completion 11-13 Years of Age vs Intervention Group: HPV Series Completion 14-17 Years of Age; Test type: Other — Chi-square tests performed to test for differences in cumulative HPV series completion vaccination rates from baseline to post-intervention; p = 0.001, Chi-squared — Statistical significance for two-sided tests was set at a type I error (alpha) equal to 0.05; Chi-square tests performed to test for differences in cumulative HPV series completion vaccination rates from baseline to post-intervention
Statistical Analysis 2: Comparison: Control Group: HPV Series Completion 11-13 Years of Age vs Control Group: HPV Series Completion 14-17 Years of Age; Test type: Other — [test comment as in outcome 2, analysis 1]; p > 0.05, Chi-squared — Statistical significance for two-sided tests was set at a type I error (alpha) equal to 0.05
Statistical Analysis 3: Comparison: Intervention Group: HPV Series Completion 11-13 Years of Age vs Control Group: HPV Series Completion 11-13 Years of Age; Test type: Other — Chi-square tests performed to test for differences in cumulative HPV series completion vaccination rates from baseline to post-intervention between intervention and control clinics; p > 0.05, Chi-squared — Statistical significance for two-sided tests was set at a type I error (alpha) equal to 0.05
Statistical Analysis 4: Comparison: Intervention Group: HPV Series Completion 14-17 Years of Age vs Control Group: HPV Series Completion 14-17 Years of Age; Test type: Other — [test comment as in outcome 2, analysis 3]; p > 0.05, Chi-squared — Statistical significance for two-sided tests was set at a type I error (alpha) equal to 0.05

ADVERSE EVENTS:
Time Frame: Baseline period to post-intervention
Arm/Group | Intervention Sites | Control Sites
Serious Adverse Events (participants affected / at risk) | 0/4942 | 0/5919
Other Adverse Events (participants affected / at risk) | 0/4942 | 0/5919

LIMITATIONS AND CAVEATS:
Limitations include: unequal distribution of baseline characteristics, possible influence of a ceiling effect, modest length (9 months) of the intervention limited ability to observe differences in HPV series completion rates between groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No